CLINICAL TRIAL: NCT05786768
Title: Efficacy and Safety of Obinutuzumab Versus Rituximab in Childhood Steroid Dependant and Frequent Relapsing Nephrotic Syndrome : a Double-blind Multicenter Randomized Controlled Study
Brief Title: Efficacy and Safety of Obinutuzumab Versus Rituximab in Childhood Steroid Dependant and Frequent Relapsing Nephrotic Syndrome
Acronym: OBIRINS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP211038; 2022-003336-59 (EudraCT Number)
Record Dates: First submitted 2023-02-10; First posted 2023-03-28 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-01

CONDITIONS: Steroid-Dependent Nephrotic Syndrome; Steroid-Sensitive Nephrotic Syndrome
Keywords: Rituximab; Obinutuzumab; Anti-Drug Antibodies
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab 375 mg/m2 (Active Comparator): single infusion of Rituximab (375 mg/m2)
  Interventions: Drug: single infusion of Rituximab
- Obinutuzumab 300 mg/1.73 m2 (Experimental): single infusion of Obinutuzumab 300 mg/1.73 m2
  Interventions: Drug: single infusion of Obinutuzumab

INTERVENTIONS:
Drug: single infusion of Rituximab — single infusion of Rituximab 375 mg/m2
  Other Names: single infusion of Rituximab 375 mg/m2
  Arms: Rituximab 375 mg/m2
Drug: single infusion of Obinutuzumab — single infusion of Obinutuzumab 300mg/1.73 m2
  Other Names: single infusion of Obinutuzumab 300mg/1.73 m2
  Arms: Obinutuzumab 300 mg/1.73 m2

SUMMARY:
B-cell depletion with rituximab induces sustained remission in children with Steroid-Dependent or Frequent Relapsing Nephrotic Syndrome (SD/FRNS). However, most patients relapse after B-cell recovery and some do not achieve B-cell depletion. Obinutuzumab is a 2nd generation humanized monoclonal antiCD20 antibody, with enhanced B cell-depleting potential. It has been reported safe and efficient in different renal autoimmune diseases including childhood nephrotic syndrome. This double-blind, randomized multicenter study is designed to assess the efficacy and safety of a single infusion of low-dose obinutuzumab compared to a single infusion of rituximab in children with frequently relapsing nephrotic syndrome (FRNS) or steroid-dependent nephrotic syndrome (SDNS).

DETAILED DESCRIPTION:
Idiopathic nephrotic syndrome (INS) is the most frequent acquired glomerulopathy in children. The initial treatment relies on steroids, which enables remission of proteinuria in 90% of children. However, 80 % of steroid-sensitive patients will relapse, and 2/3 will become steroid-dependant with a long lasting disease over years. In this situation, immunosuppressive drugs are added as steroid-sparing agents. There is no international consensus on the second line treatment strategy after initial steroid therapy. RCT have demonstrated the efficacy of rituximab (RTX) to maintain remission in FR/SDNS after oral treatments withdrawal, however most patients relapse within 2 years, and some patients are resistant or allergic to Rituximab. Obinutuzumab (OBI) is a second generation antiCD20 mAb, that has been designed to overcome rituximab resistance in B-cell malignancies. Additional mechanisms of rituximab failure support the hypothesis that B-cell depletion could be optimized with OBI in autoimmune diseases. OBI has met its primary endpoint in lupus nephritis and a few randomized controlled trials are currently ongoing in nephrology for lupus nephritis and membranous nephropathy. We believe that a single infusion of OBI could reduce the risk of subsequent relapse in FR/SDNS and the cumulative exposure to immunosuppressive drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 18 years
* Steroid dependant Nephrotic Syndrome defined as:

  * 2 or more relapses during steroids or within 2 weeks following discontinuation.
  * 2 or more relapses including one under steroid-sparing agent (MMF, Calcineurin inhibitors, cyclophosphamide, levamisole) or within 6 months following treatment withdrawal

OR Frequent Relapsing Nephrotic Syndrome defined as:

* 2 or more relapses within 6 months following first remission
* 3 or more relapses within any 12-month period

  * Last relapse within 3 months prior to inclusion
  * In remission, defined as 3 consecutive urinary dipsticks without proteinuria, at the time of randomization
  * Vaccination schedule in accordance with the current recommendations in France
  * Informed consent from parents

Exclusion Criteria:

* Secondary cause of nephrotic syndrome (such as membranous nephropathy, IgA nephropathy, lupus nephritis)
* Primary or secondary steroid resistance nephrotic syndrome
* Prior treatment with Rituximab within 6 months
* Prior treatment with obinutuzumab at any time
* CD20+ B-cell count < 2.5%
* Patient with neutrophils < 1.5 G/L and/or platelets < 75 G/L
* GFR < 80 ml/min/1.73m2
* Weight <16kg
* History of severe infection such as tuberculosis, hepatitis B, hepatitis C or HIV infection or LEMP
* History of malignancy- Uncontrolled infection (viral, bacterial and fungal)
* Vaccination with a live vaccine within 4 weeks prior to assignment/randomization
* Known hyperprolinemia
* Hypersensitivity to the active substance (OBI or RTX) or to proteins of murine origin, or to any of the other excipients
* Pregnancy or breastfeeding or ability to become pregnant and refusal to use effective contraception during the 18 months following the study treatment (only 1 infusion of obinutuzumab/Rituximab at the beginning of the study)
* Patient without medical insurance coverage (beneficiary or legal)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2027-10-18 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a relapse within 12 months following the initiation of treatment | 12 months
  Relapse is defined as a protein to creatinine ratio of 2 g/g of creatinine (0.20 g/mmol) or higher

SECONDARY OUTCOMES:
Occurrence of a relapse within 24 months | 24 months
Time to B-cell depletion | 24 months
Duration of relapse-free survival after B-cell reconstitution | 24 months
Cumulative steroid courses and second line immunosuppressive treatments in patients with relape | 24 months
Safety associated with drug infusion | 24 months
  Nature, frequency and timing of side effects
Efficiency defined as incremental cost-effectiveness ratio in cost per relapse prevented | 24 months
Budgetary impact defined as costs and health gains incurred with the generalization of the obinutuzumab strategy | 24 months
Detection of Antidrug Antibodies | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Claire DOSSIER, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 48 months

REFERENCES:
- [Derived] Dossier C, Sellier-Leclerc AL, Simon T, Parmentier C, Boyer O, Samaille C, Fila M, Roussey-Kesler G, Magnavacca M, Chartier Y, Louillet F, Zaloszyc A, Vrillon I, Elaribi D, Bouatia S, Kaguelidou F, Guilmin-Crepon S, Hogan J. Obinutuzumab versus Rituximab to maintain remission in children with steroid-dependent and frequently relapsing nephrotic syndrome: the OBIRINS study protocol, a double-blind randomised controlled trial. BMJ Open. 2025 Dec 24;15(12):e111980. doi: 10.1136/bmjopen-2025-111980. PMID 41448676
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526
- [Derived] Dossier C, Bonneric S, Baudouin V, Kwon T, Prim B, Cambier A, Couderc A, Moreau C, Deschenes G, Hogan J. Obinutuzumab in Frequently Relapsing and Steroid-Dependent Nephrotic Syndrome in Children. Clin J Am Soc Nephrol. 2023 Dec 1;18(12):1555-1562. doi: 10.2215/CJN.0000000000000288. Epub 2023 Sep 6. PMID 37678236